CLINICAL TRIAL: NCT02273466
Title: Pharmacokinetics of 50 mg Desipramine Daily, Given Orally Over 7 Days With and Without Concomitant Administration of 175 mg Crobenetine, Given as a 6 Hrs i.v. Infusion (One Hour Loading Dose Directly Followed by a Five Hours Maintenance Dose). A Randomized, Placebo Controlled, Single Blind (for Crobenetine), Two-way Cross Over Trial in Healthy Male Subjects
Brief Title: Pharmacokinetics of Oral Desipramine With and Without Concomitant Administration of Crobenetine Infusion in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 599.11
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Desipramine

ARMS (2):
- Desipramine alone (Active Comparator)
  Interventions: Drug: Desipramine tablet; Drug: Placebo infusion
- Desipramine with Crobenetine (Experimental)
  Interventions: Drug: Desipramine tablet; Drug: Crobenetine infusion

INTERVENTIONS:
Drug: Desipramine tablet
Drug: Crobenetine infusion
  Arms: Desipramine with Crobenetine
Drug: Placebo infusion
  Arms: Desipramine alone

SUMMARY:
To assess the steady state pharmacokinetics of Desipramine with/without concomitant administration of Crobenetine.

ELIGIBILITY:
Inclusion Criteria:

All participants in the study should be healthy males, range from 21 to 50 years of age and their bodymass index (BMI) be within 18.5 to 29.9 kg/m2.

In accordance with Good Clinical Practice and local legislation all volunteers will have given their written informed consent prior to admission to the study.

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial (within one week prior to administration or during the trial)
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (>= 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range of clinical relevance
* Cytochrome P450 2D6 poor metaboliser (to be determined by phenotyping or genotyping)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-02; Primary Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve for desipramine at steady state (AUC,ss) | up to 168 hours after start of drug administration
Maximum plasma concentration of desipramine at steady state (Cmax,ss) | up to 168 hours after start of drug administration

SECONDARY OUTCOMES:
Individual time courses of plasma concentrations | up to 168 hours after start of drug administration
Area under the concentration time curve from zero time to time of last quantifiable drug concentration (AUC0-tz) | up to 168 hours after start of drug administration
Area under the concentration time curve from zero time extrapolated to infinity(AUC0-infinity) | up to 168 hours after start of drug administration
Time to reach maximum concentration of desipramine at steady state (tmax,ss) | up to 168 hours after start of drug administration
Apparent terminal rate constant (λz) | up to 168 hours after start of drug administration
Apparent terminal half-live in plasma (t1/2) | up to 168 hours after start of drug administration
Mean residence time (MRT) | up to 168 hours after start of drug administration
Total clearance (CL) | up to 168 hours after start of drug administration
Apparent volume of distribution (V) | up to 168 hours after start of drug administration
Observed concentration of crobenetine (C,h) | 1 and 6 hours after start of infusion
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with clinically significant findings in vital signs | up to 8 days after last drug administration
  blood pressure, pulse rate
Number of subjects with clinically significant findings in 12-lead ECG | up to 8 days after last drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 8 days after last drug administration